CLINICAL TRIAL: NCT06275581
Title: Clinical Evaluation of the Performance of a Newly Developed Glass Ionomer Restorative for Posterior Restorations in an Adult Population: Pilot Study
Brief Title: Clinical Evaluation of the Performance of a Newly Developed Glass Ionomer Restorative for Posterior Restorations in an Adult Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR15_15 (EM-11-050055)
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Tooth Wear; Glass Ionomer Cements
Keywords: tooth wear; dental restoration; dental impression
MeSH Terms: conditions — Tooth Wear | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketac Universal test group (Experimental): intra-individual (split-mouth) study
  Interventions: Device: Ketac Universal Aplicap Glass Ionomer Restorative (3M) (test group)
- Ketac Molar Quick control group (Active Comparator): intra-individual (split-mouth) study
  Interventions: Device: Ketac Molar Quick Aplicap Glass Ionomer Restorative (control group)

INTERVENTIONS:
Device: Ketac Universal Aplicap Glass Ionomer Restorative (3M) (test group) — Ketac Universal Aplicap Glass Ionomer Restorative (test group) was applied in one cavity of the patient, randomized allocated, in a stress bearing Class II restoration when the isthmus was less than half of the intercuspal distance and with at least one occlusal contact on enamel of the restored tooth. This material does not require a cavity conditioning step prior to restoration placement.
  Arms: Ketac Universal test group
Device: Ketac Molar Quick Aplicap Glass Ionomer Restorative (control group) — Ketac Molar Quick Aplicap Glass Ionomer Restorative (control group) was applied in the other cavity of the patient,randomized allocated, in a stress bearing Class II restoration when the isthmus was less than half of the intercuspal distance and with at least one occlusal contact on enamel of the restored tooth.
  Arms: Ketac Molar Quick control group

SUMMARY:
STUDY DESIGN Post market clinical follow-up; pilot study, prospective, controlled, randomized, split-mouth, blinded evaluation INTRODUCTION AND PURPOSE OF STUDY Continuous advancements in the field of glass ionomers have led to an increasing range of permanent indications, especially with regards to stress bearing Class II restorations. As a further development in the 3M glass ionomer category, Ketac Universal can be used for the abovementioned indication in a simplified procedure without the need for cavity conditioning or restoration coating. All products used in this study are CE marked thus can be used for routine clinical treatment.

STUDY OBJECTIVES Objective of the study is to evaluate the clinical survival and quality parameters of Class II Ketac Universal restorations compared to intra-individual (split-mouth) Class II Ketac Molar Quick control restorations over time STUDY ENDPOINTS

Primary Endpoint:

1. Evaluation of restoration survival over time based on the glass ionomer restoration criteria (simplified FDI criteria as proposed by Mathilde Peters et al.)

Secondary Endpoints:

1. Evaluation of restoration quality based on the glass ionomer restoration criteria (simplified FDI criteria)
2. Evaluation of restoration wear based on comparison of digital impressions

Safety Endpoint:

1. Evaluation of potential adverse events NULL HYPOTHESIS There is no statistically significant difference between both glass ionomers

* regarding overall survival
* regarding restoration quality parameters TEST GROUP Ketac Universal Aplicap Glass Ionomer Restorative (3M) CONTROL GROUP Ketac Molar Quick Aplicap Glass Ionomer Restorative (3M)
* regarding restoration wear METHODS AND MATERIALS A total of 39 subjects were enrolled and treated. The study was originally planned with 80 patients. Due to slow recruitment, it was decided to decrease the number of patients.

Treatment:

After signing informed consent, test and control product were randomly assigned to the two study teeth (randomization letter). Restoration extension (e.g. mod) and reason for restoration placement (e.g. secondary caries, tooth fracture) were recorded in the CRF. Two teeth per subject were included. Each product was used strictly according to respective Instructions for Use without using the optional protective coating. Restorations were placed in combination with sectional matrix system (Palodent system) and according to best practice (especially with regards to moisture control). Finishing and polishing was done with the Sof-Lex system. Areas in close proximity to the pulp were covered with local application of a calcium hydroxide material in both study materials. Study teeth were excluded from study if pulp exposure had occurred or if only a repair restoration was required instead of a full Class II restoration.

Evaluation periods:

All subjects were evaluated by two independent evaluators according to Performance Criteria for Posterior Glass Ionomer Restorations (simplified FDI criteria)

* at baseline at day of restoration placement or up to 1 month after restoration placement
* after 6 months (± 1 months)
* after 1 year (± 1 months)
* after 2 years (± 1 months) In addition, photos (at least occlusal view) were taken of every study tooth prior to restoration placement and at every evaluation.

In order to further assess the wear of both restorative materials, full arch digital impressions (both upper and lower jaw) were taken at baseline evaluation and at every following evaluation using 3M True Definition Scanner. STL files were digitally compared to those taken at baseline.

DETAILED DESCRIPTION:
INTRODUCTION First generation glass ionomers were introduced into the market in the early 1970ies. In the beginning glass ionomers were indicated only for temporary restorations or non-stress bearing restorations of limited size. Continuous advancements of the glass ionomer chemistry have led to an increasing range of permanent indications, especially with regards to stress bearing Class II restorations.

Ketac Molar Quick, the control material used in this clinical study, is indicated for such stress bearing restorations, but still requires a mandatory conditioning step prior to restoration placement. As a further development in the 3M glass ionomer category, Ketac Universal can be used for the abovementioned indication in a simplified procedure without the need for cavity conditioning.

The aim of the present investigation is to evaluate the clinical survival and development of quality parameters of Class II restorations using Ketac Universal over time. As a control, Ketac Molar Quick Class II restorations are placed in a split-mouth design.

4.0 METHODS 4.1 Study Device Information Both Ketac Universal and the control material Ketac Molar Quick are glass ionomer restoratives with almost identical range of indications (including, but not limited to, stress bearing Class II restorations when the isthmus is less than half of the intercuspal distance and with at least one occlusal contact on enamel of the restored tooth). Both materials have been used in commercially available CE marked dosage form and have been used according to Instructions for Use without the optional protective coating step.

The difference between Ketac Universal and Ketac Molar Quick is that Ketac Universal has a softer consistency and does not require a cavity conditioning step prior to restoration placement.

4.1.1 Test group Test group: 3M KETAC TM UNIVERSAL APLICAP GLASS IONOMER RESTORATIVE This product is commercially available, bears the CE sign and can therefore be used for routine clinical treatment.

KetacTM Universal AplicapTM is a radiopaque glass ionomer restorative in capsules used for bulk fillings. The ability of the material to bond chemically to enamel and dentin ensures gentle preparation and excellent sealing on the margins of fillings. Ketac Universal Aplicap can be applied without lining; it releases fluoride ions and is available in various shades corresponding to the VitaTM Classical color system. The dispensable quantity of a capsule is at minimum 0.13 ml.

4.1.2 Control Group In the control group, 3M KETAC TM MOLAR Quick Aplicap Glass Ionomer Restorative was used. This product is commercially available, bears the CE sign and can therefore be used for routine clinical treatment.

KetacTM Molar Quick AplicapTM is a glass ionomer cement in a capsule. On account of its chemical adhesion to the dental enamel and dentin, a gentle preparation and an especially tight seal at the margins is possible. The product is available in the following shades: A1, A2, A3, A4 and B2. The material can be applied without lining; it releases fluoride ions and is radiopaque. The dispensable quantity of a capsule is at least 0.13 ml.

Additional 3M material not in focus of this study was used in the dental procedures.

4.2 Study Objectives and Endpoints The objective of the study is to evaluate the clinical survival and quality parameters of Class II test restorations compared to intra-individual (split-mouth) Class II control restorations over time.

The null hypothesis is that the clinical performance of test and control restorations is similar regarding all endpoints.

4.2.1 Primary Endpoint: The primary endpoint in this study is the evaluation of restoration survival over time based on the glass ionomer restoration criteria . Restoration survival is defined as following: A restoration is classified as "survival" if it has received score 1 through 3 in all categories. In case of non-acceptable performance (score 4 or score 5 in one or more of the glass ionomer restoration criteria (simplified FDI criteria) the restoration is classified as a failure.

4.2.2 Secondary Endpoints: Two secondary endpoints are evaluated in this study.

1. Evaluation of restoration quality based on the glass ionomer restoration criteria (Individual restauration performance (score 1 through 5) in each category according to glass ionomer restoration criteria
2. Evaluation of restoration wear based on comparison of digital impressions 4.2.3 Safety Endpoint: The safety endpoint is the incidence of Adverse Events. 4.3 Description of Study Design and Plan 4.3.1 Selection of Study Population 57 subjects were assessed for eligibility during routine intraoral examinations. 18 did not meet the inclusion criteria. After obtaining written informed consent a total of 39 adult patients were initially selected for the study after identification during routine clinical examinations. 3 of the 39 patients were excluded as they only required repair of already existing, defective fillings instead of full Class II restorations, so the total population of the study is 36 patients. Originally, it was planned to treat 80 patients. Due to slow recruitment it was decided to decrease the number of patients.

Inclusion and Exclusion criteria are listed in the table below.

4.3.3 Study Design This study is a post market clinical follow-up study with CE marked products used per label. The study design is prospective, randomized, controlled, split-mouth, independent and blinded evaluation.

Originally, the study was planned for 5 years follow-up. However, due to the Covid-19 pandemic and the associated drop-out rate it was decided to terminate the study with data available until January 2021.

Start of study Screening of patients for inclusion/exclusion criteria, mainly: in need of Class II restorations on 2 teeth with good prognosis for the next 5 years Signing of informed consent & enrollment of 80 adult subjects into the study Restoration placement Randomized allocation of treatment to the 2 study teeth according to randomization list; photo documentation of study teeth prior to treatment Assignment of Ketac Universal to one study tooth Assignment of Ketac Molar with Conditioner to the other study tooth Placement of Class II restorations according to assignment in combination with sectional matrix system and according to best practice (especially with regards to moisture control); finishing and polishing with the Sof-Lex system; no placement of optional protective coat; cover areas in close proximity to the pulp with local application of a calcium hydroxide material; Exclude tooth if pulp exposure has occured T0 Baseline evaluation + Full arch digital impression + Photo at day of restoration placement or up to 1 month after restoration placement by two independent blinded evaluators according to evaluation criteria T6MONTHS Evaluation + Full arch digital impression + Photo 6 months (±1 month) after restoration placement by two independent blinded evaluators according to evaluation criteria T1 Evaluation + Full arch digital impression + Photo 1 year (±1 month) after restoration placement by two independent blinded evaluators according to evaluation criteria T2 Evaluation + Full arch digital impression + Photo 2 years (±1 month) after restoration placement by two independent blinded evaluators according to evaluation criteria

4.3.4 Treatment and Evaluation Patients were recruited in the Department of Prosthodontics after identification during routine clinical examinations. Study started on 2017-06-14 with the first patient in, and it ended on 2021-03-24 with last patient out.

After signing informed consent, test (Ketac Universal) and control product (Ketac Molar Quick) were randomly assigned to the two study teeth per randomization letter. If a subject was in need of more than 2 Class II restorations, the two most comparable Class II restorations were included (based on restoration size). Additional teeth requiring treatment were not be part of the study and were treated according to clinical routine.

Restoration extension (e.g. mod) and reason for restoration placement (e.g. secondary caries, tooth fracture) were recorded on the CRFs. Only two teeth per subject were included.

For details on placement procedure please refer to the respective Instructions for Use. Main difference between Ketac Universal and Ketac Molar Quick placement is that Ketac Molar Quick requires a cavity conditioning step before placement while Ketac Universal does not. The restorations were placed in bulk-fill mode.

Teeth were cleaned to remove surface stains. Prior to isolation of teeth, the appropriate shade(s) of Ketac Universal and Ketac Molar were selected using a standard VITAPAN® classical shade guide.

Restoration placement was done according to best practice (e.g. proper working field isolation) and in combination with a sectional matrix system (Palodent system). All restorations were finished and polished with the Sof-Lex system. Restorations did not receive the optional protective coating. Areas in close proximity to the pulp were covered with local application of a calcium hydroxide material in both materials; study teeth were excluded if a pulp exposure had occurred.

Blinding of operators was not feasible due to application differences between both study materials. Ketac Molar Quick requires a conditioner while Ketac Universal does not. Evaluators were blinded with regard to restoration material used. Blinding during evaluation was possible because the esthetic appearance of Ketac Universal and Ketac Molar Quick is very similar.

All Class II restorations needed to fulfill the following criteria: located in a stress bearing area and in addition at least one occlusal contact on enamel of restored tooth, isthmus (if present) less than half of intercuspal distance, restoration must have proximal contact, no cusp replacement.

All subjects were evaluated by two independent evaluators according to Performance Criteria for Posterior Glass Ionomer Restorations (simplified FDI criteria) at the following time points:

* at baseline at day of restoration placement or up to 1 month after restoration placement
* after 6 months (± 1 months)
* after 1 year (± 1 months)
* after 2 years (± 1 months) In addition, photos (at least occlusal view) were taken of every study tooth prior to restoration placement and at every evaluation.

In order to further assess wear of both restorative materials, full arch digital impressions (both upper and lower jaw) were taken at baseline evaluation and at every following evaluation using 3M True Definition Scanner. STL files at each evaluation were digitally compared to those taken at baseline.

The recall visits included a free full mouth revision and cleaning. At restoration placement the restored surfaces and additional info were documented in the CRF and the respective FDI tooth number.

Following criteria were evaluated for study teeth individually by two evaluators and their consensus (Clinical Performance Criteria for Posterior Glass Ionomer Restorations (simplified FDI criteria)):

* Retention
* Fractures / Marginal Chipping
* Surface / Marginal Staining
* Wear
* Postoperative Sensitivity / Vitality
* Caries Associated with Restoration (CAR)
* Tooth Integrity (enamel cracks / tooth fracture)

4.4 Statistical Methods of Analysis 4.4.1 Sample Size Determination In the initial study protocol, it was intended to enroll 80 patients, with an estimated 30% drop-out rate. This sample size exceeds the requirements of the ADA Acceptance Program Guidelines "Tooth-Colored Restorative Materials for Posterior Teeth" which requires a minimum of 40 restorations in 20 patients. Due to slow recruitment, the target was decreased to 39 patients per protocol amendment, still exceeding ADA patient number requirements.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 70 years of age
* Subject is in good general health
* Subject does not have known allergies against any study substances
* Subject is in need of a Class II restoration on at least 2 teeth (stress bearing, isthmus less than half of intercuspal distance, no cusp replacement)
* Both study teeth must have a good prognosis for the next 5 years (no increased tooth mobility, periodontal probing depth is ≤5 mm, no signs of pulpitis, no pulp exposure during treatment, tooth is vital, level of oral hygiene is sufficient)
* Both study restorations are not in contact to each other
* Subject does not suffer from bruxism or from traumatic malocclusion
* Study tooth must have one enamel supported antagonistic contact outside the restoration area
* Each study restoration has at least one proximal contact and is stress bearing
* Subject does not have excessive dietary or environmental exposure to acids or suffer from eating disorders
* Subject is not pregnant or breast feeding
* Subject volunteers to participate in the study and is available for recalls during the 5 years study duration
* Subject does not participate in any other study

Exclusion Criteria:

-

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Restoration survival over time based on the glass ionomer restoration criteria | 1-24 months
  Restoration survival is defined as following: A restoration is classified as "survival" if it has received score 1 through 3 in all categories. In case of non-acceptable performance (score 4 or score 5 in one or more of the glass ionomer restoration criteria -simplified FDI criteria- the restoration is classified as a failure.
  The Clinical Performance Criteria for Posterior Glass Ionomer Restorations -simplified FDI criteria- scores the following aspects:
  Retention, Fractures / Marginal Chipping, Surface / Marginal Staining, Wear, Postoperative Sensitivity / Vitality, Caries Associated with Restoration (CAR), Tooth Integrity (enamel cracks / tooth fracture).
  The Evaluation periods for the FDI criteria were:
  at baseline at day of restoration placement or up to 1 month after restoration placement, after 6 months (± 1 months), after 1 year (± 1 months), after 2 years (± 1 months).

SECONDARY OUTCOMES:
Evaluation of restoration quality based on the glass ionomer restoration criteria | 1-24 months
  Individual restoration performance (score 1 through 5) in each category according to glass ionomer restoration criteria. This simplified FDI criteria analyzes: Retention, Fractures / Marginal Chipping, Surface / Marginal Staining, Wear, Postoperative Sensitivity / Vitality, Caries Associated with Restoration (CAR), Tooth Integrity (enamel cracks / tooth fracture).
Evaluation of restoration wear based on comparison of digital impressions | 1-24 months
  True Definition intraoral scanner was used to scan the restorations at each of the evaluation periods. The STL files obtained by those optical impressions were superimposed and compared.
Safety Endpoint: The safety endpoint is the incidence of Adverse Events. | 1-24months
  To report any adverse events if happen

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Health Clinic at Universidad Europea de Madrid (UEM) Department of Prosthodontics, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urcelay Moreno N, Bertuol Gessi SF, Benabdallah M'Rabat M, Thuissard IJ, Santamaria-Laorden A. In vivo prospective randomised study of the wear of dental restorations using an intraoral scanner and its correlation with visual assessment. J Dent. 2025 Feb;153:105471. doi: 10.1016/j.jdent.2024.105471. Epub 2024 Nov 26. PMID 39603331